CLINICAL TRIAL: NCT04174014
Title: Estimation of Optimal PEEP by Transpulmonary Pressure Measurement Following Recruitment Manoeuvre Under Computer Tomography and Electric Impedance Tomography Control
Brief Title: Optimal PEEP Titration Combining Transpulmonary Pressure Measurement and Electric Impedance Tomography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kiskunhalas Semmelweis Hospital the Teaching Hospital of the University of Szeged (Other Government)
Collaborators: Budapest University of Technology and Economics (Other); Hochschule Furtwangen University (Other); Szeged University (Other)
Responsible Party: Principal Investigator, András Lovas, MD, PhD, EDIC, EDAIC, head of department, Kiskunhalas Semmelweis Hospital the Teaching Hospital of the University of Szeged
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTP
Record Dates: First submitted 2019-11-03; First posted 2019-11-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recruitment manoeuvre (Experimental): 1. Volume control (VC) ventilation mode with a tidal volume of 6 mL/kg of ideal body weight
  2. P/V tool assessment
  3. Baseline measurements
  4. CT scan of chest without EIT belt
  5. Re-establishment of EIT belt, continuous EIT and transpulmonary pressure measurement during the recruitment and de-recruitment manoeuvre.
     increment phase:
     * constant volume settings
     * increasing PEEP with 4 cmH2O following each 10 consecutive controlled breath until reaching a peak pressure of 40 cmH2O
     decrement phase:
     * constant volume settings
     * decreasing PEEP with 4 cmH2O following each 10 consecutive controlled breath not lower than 2 cmH20 from target PEEP
     * target PEEP level is defined where the end-expiratory transpulmonary pressure is 0-1 cmH2O
  6. P/V recruitment with target end-PEEP level
  7. Removal of EIT belt, CT scan of chest
  8. Continuous EIT and transpulmonary pressure measurement with the initial FiO2 and the new PEEP settings
  Interventions: Procedure: Recruitment manoeuvre

INTERVENTIONS:
Procedure: Recruitment manoeuvre — PEEP increment and decrement

SUMMARY:
Diagnosis and treatment of the hypoxic respiratory failure induced by severe atelectasis with the background of acute lung injury is challenging for the intensive care physicians. Mechanical ventilation commenced with grave hypoxemia is one of the most common organ support therapies applied in the critically ill. However, respiratory therapy can improve gas exchange until the elimination of the damaging pathomechanism and the regeneration of the lung tissue, mechanical ventilation is a double edge sword. Mechanical ventilation induced volu- and barotrauma with the cyclic shearing forces can evoke further lung injury on its own.

Computer tomography (CT) of the chest is still the gold standard in the diagnostic protocols of the hypoxemic respiratory failure. However, CT can reveal scans not just about the whole bilateral lung parenchyma but also about the mediastinal organs, it requires the transportation of the critically ill and exposes the patient to extra radiation. At the same time the reproducibility of the CT is poor and it offers just a snapshot about the ongoing progression of the disease. On the contrary electric impedance tomography (EIT) provides a real time, dynamic and easily reproducible information about one lung segment at the bed side. At the same time these picture imaging techniques are supplemented by the pressure parameters and lung mechanical properties assigned and displayed by the ventilator. The latter can be ameliorated by the measurement of the intrapleural pressure. Through with this extra information transpulmonary pressure can be estimated what directly effects the alveoli.

Unfortunately, parameters measured by the respirator provide only a global status about the state of the lungs. On the contrary acute lung injury is characterized by focal injuries of the lung parenchyma where undamaged alveoli take part in the gas exchange next to the impaired ones. EIT can aim the identification of these lesions by the assessment of the focal mechanical properties when parameters measured by the ventilator are also involved. The latter one can not just take a role in the diagnosis but with the support of it the effectivity of the alveolar recruitment can be estimated and optimal ventilator parameters can be determined preventing further damage caused by the mechanical stress.

DETAILED DESCRIPTION:
Following PEEP increment and decrement alveolar recruitment manoeuvre optimal PEEP would be assessed by transpulmonary pressure measurement to keep open up the lung. Physicians are lack of data at which pressure the most alveoli are recruited and if 40 cmH2O of pressure is really required for complete recruitment. By CT scan of chest and continuous EIT measurement rate of recruitment would be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Orotracheally intubated patients ventilated in volume control mode with moderate and severe hypoxic respiratory failure according to the ARDS Berlin definition.
* 100 Hgmm ≤ PaO2/FiO2 ≤ 200 Hgmm, PEEP ≥ 5 cmH2O (moderate) or PaO2/FiO2 ≤ 100 Hgmm, PEEP ≥ 5 cmH2O (sever)

Exclusion Criteria:

* age under 18
* pregnancy
* pulmonectomy, lung resection in the past medical history
* clinically end stage COPD
* sever hemodynamic instability (vasopressor refractory shock)
* sever bullous emphysema and/or spontaneous pneumothorax in the past medical history
* chest drainage in situ due to pneumothorax and/or bronchopleural fistula
* contraindication of the application of oesophageal balloon catheter (oesophageal ulcer, oesophageal perforation, oesophageal diverticulosis, oesophageal cancer, oesophageal varices, recent operation on oesophagus and/or stomach, sever coagulopathy)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Highest level of transpulmonary pressure to open up the lung | 1 minute
  Estimation of the highest level of transpulmonary pressure (cmH2O) during the increment PEEP phase when the end-expiratory lung volume (ml) can not be increased further
Changes between the two PEEP level (titrated by transpulmonary pressure measurement vs. optimal PEEP by EIT) estimated in cmH2O control | 15 minutes
  PEEP settings by keeping the transpulmonary pressure around 1 cmH2O at an end-expiratory hold manoeuvre really represents the most optimal circumstances by electric impedance tomography as well. Optimal circumstances by EIT would be represented by at the crossover point of hyperdistension/collapse % curves plotted versus PEEP. Difference between the two PEEP level (titrated by transpulmonary pressure measurement vs. optimal PEEP by EIT described previously) would be estimated (cmH2O).

SECONDARY OUTCOMES:
Gas exchange | 30 minutes
  Change in PaO2 (mmHg) following recruitment
Plateau pressure | 30 minutes
  Change in plateau pressure (cmH2O) under volume control ventilation mode
Transpulmonary pressure | 30 minutes
  Change in transpulmonary pressure (cmH2O) following intervention
Estimation in recruitability | 30 minutes
  Change in end expiratory lung volume (ml) following intervention
Antero-to-posterior ventilation ratio | 30 minutes
  Change in antero-to-posterior ventilation ratio (%) following intervention
Center of ventilation | 30 minutes
  Change in center of ventilation (%) following intervention
Global inhomogeneity index | 30 minutes
  Change in global inhomogeneity index (%) following intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Department of Anesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chiumello D, Brochard L, Marini JJ, Slutsky AS, Mancebo J, Ranieri VM, Thompson BT, Papazian L, Schultz MJ, Amato M, Gattinoni L, Mercat A, Pesenti A, Talmor D, Vincent JL. Respiratory support in patients with acute respiratory distress syndrome: an expert opinion. Crit Care. 2017 Sep 12;21(1):240. doi: 10.1186/s13054-017-1820-0. PMID 28899408
- [Result] Marini JJ. Evolving concepts for safer ventilation. Crit Care. 2019 Jun 14;23(Suppl 1):114. doi: 10.1186/s13054-019-2406-9. PMID 31200734
- [Result] Pesenti A, Musch G, Lichtenstein D, Mojoli F, Amato MBP, Cinnella G, Gattinoni L, Quintel M. Imaging in acute respiratory distress syndrome. Intensive Care Med. 2016 May;42(5):686-698. doi: 10.1007/s00134-016-4328-1. Epub 2016 Mar 31. PMID 27033882
- [Result] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Result] Yoshida T, Brochard L. Esophageal pressure monitoring: why, when and how? Curr Opin Crit Care. 2018 Jun;24(3):216-222. doi: 10.1097/MCC.0000000000000494. PMID 29601320
- [Result] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Result] Lovas A, Szakmany T. Haemodynamic Effects of Lung Recruitment Manoeuvres. Biomed Res Int. 2015;2015:478970. doi: 10.1155/2015/478970. Epub 2015 Nov 22. PMID 26682219